CLINICAL TRIAL: NCT04447677
Title: Correlation of Progesterone Levels on the Day of Oocyte Retrieval With Basal Hormonal Status and the Outcome of in Vitro Fertilization in Women
Brief Title: Oocyte Retrieval Progesterone Levels and IVF
Status: Completed | Type: Observational
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Lidija Tulic, Assistent Professor, University of Belgrade
Other Study IDs: 25138
Record Dates: First submitted 2020-06-11; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Hormone Disturbance
MeSH Terms: conditions — Endocrine System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
Objective: To assess whether basal hormonal level can predict the elevation of P4 on the day of oocyte retrieval, as well as to examine the impact of P4 elevation on the day of oocyte retrieval on the outcome of assisted reproduction.

Design: Prospective cohort study Setting: Department of In Vitro Fertilization, Gynecology and Obstetrics Institute, Clinical Center of Serbia Patient(s): One hundred sixty four patients enrolled in the ART procedure Main Outcome Measure(s): Pregnancies, miscarriages, biochemical pregnancies and deliveries

DETAILED DESCRIPTION:
A prospective clinical trial was conducted at the Clinic for Gynecology and Obstetrics Clinical Center of Serbia from January 1st to December 31st 2015. The study included 164 patients enrolled in the ART procedure at the Clinic.

Basal hormonal status - serum levels of estradiol (E2 - pg/ml), progesterone (P4 - ng/ml), follicle-stimulating hormone (FSH - mIU/ml), luteinizing hormone (LH - mIU/ml) and anti-Mullerian hormone (AMH - ng/l) were measured on the 2ndor 3rd cycle day before stimulation commencement. During COS levels of estradiol were determined, while levels of progesterone were determined on the day of oocyte retrieval i.e. aspiration. Blood samples were taken by Vacutainer tubes (BD Vacutainer Systems) and centrifuged according to the manufacturer's instructions for the preparation of the serum samples. AMH value (Gen II ELISA ref. No. A79765; Beckman Coulter) in serum was measured by ELISA (enzyme-linked immunosorbent assay), 1 ng / ml). FSH, LH, estradiol, and progesterone were analyzed by chemiluminescent immunoassay (Access 2 immunoassay system, Beckman Coulter).

The main outcome measures were the procedure success as well as the pregnancy outcome. Pregnancy was confirmed by a positive finding of serum β-hCG (>25 MIU/ml) 14 days after embryo transfer. Clinical pregnancies were confirmed by transvaginal ultrasound findings of a gestational sac with a vital embryo at the 6th gestational week.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years of age
* BMI of 18 to 30 kg/m2
* regular menstrual cycles from 25 to 32 days
* established diagnosis of infertility.

Exclusion Criteria:

* Less then 18 or more then 40 years old
* BMI less then 18 or more then 30 kg/m2
* irregular menstrual cycles

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study evaluated 164 patients undergoing ART procedure - oocyte retrieval and embryo transfer in our Clinic. Patients in average had 34.66 ± 3.39 years, mean BMI was 22.23 ± 2.65, and their infertility mostly lasted for 4.86 ± 2.61 years (range 1 to 17 years).
  The mean P4 values on OR day were 1.26 ± 0.46 ng/ml in group P4 <2ng/ml, while in the group of patients with P4 values ≥2ng/ml, the average P4 was 3.74 ± 1.62 ng/ml.
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Outcome of Ivf procedure | 12 months
  Outcome of ivf procedure can be positive and devided in pregnancies, miscariages or biochemical pregnancies or can be negative outcome -failire of procedure

IPD SHARING:
Plan to Share IPD: Undecided